CLINICAL TRIAL: NCT04093947
Title: Characteristics of Subjects With Overweight or Obesity at the Onset of Hypertension
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Gianluigi Giannelli, Clinical Professor, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: prot2019
Record Dates: First submitted 2019-08-27; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Hypertension; Obesity
MeSH Terms: conditions — Hypertension; Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Observational and prospective study

SUMMARY:
The study aims to investigate the characteristics of subjects with hypertension at onset among a cohort of apparently healthy subjects, with overweight or obesity (BMI ≥ 25 Kg / m2), and free of any drug treatment at the baseline. The evaluation includes anthropometric (weight, height, BMI, waist circumference), haematochemical (hormones, metabolic and routine) parameters and the screening for hypertension with ABPM. The diagnosis of hypertension is made in accordance with the 2017 guidelines of the American College of Cardiology / American Heart Association ACC / AHA.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI> 25 Kg/m2)

Exclusion Criteria:

* Any kind of drug
* Hypertension
* Endocrine diseases (diabetes mellitus, hypo or hyperthyroidism, hypopituitarism, etc.),
* Chronic inflammatory diseases
* Renal failure
* Liver failure
* Angina pectoris
* Myocardial infarction and heart failure
* Genetic heart diseases
* Thrombocytopenias

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who came to the Outpatient Clinic of Nutrition at the National Institute of Gastroenterology "S. de Bellis," Research Hospital, Castellana Grotte, Italy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Insulin | At baseline
  Insulin (mIU/L) concentration in serum
Potassium | At baseline
  Potassium (mmol/L) concentration in serum
Sodium | At baseline
  Sodium (mEq/L) concentration in serum
eGFR (estimated glomerular filtration rate) | At baseline
  eGFR (ml/min/1.73 mq)
Creatinin | At baseline
  Creatinin (mg/dl) concentration in serum
Uric acid | At baseline
  Uric acid (mg/dL) concentration in serum
Total cholesterol | At baseline
  Total cholesterol (mg/dL) concentrations in serum
Thyroid hormones (FT3, FT4) | At baseline
  FT3 (pg/mL), FT4 (pg/mL) concentration in serum
HDL cholesterol | At baseline
  HDL cholesterol (mg/dL) concentrations in serum
LDL cholesterol | At baseline
  LDL cholesterol (mg/dL) concentrations in serum
Triglycerides | At baseline
  Triglycerides (mg/dL) concentrations in serum
TSH | At baseline
  TSH (mU/L) concentration in serum

SECONDARY OUTCOMES:
BMI | At baseline
  BMI (kg/m^2)
Height | At baseline
  Height in meters
Weight | At baseline
  Weight in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Gastroenterology IRCCS S. de Bellis, Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No